CLINICAL TRIAL: NCT01140737
Title: A Clinicopathological Phase II Study of Axitinib in Patients With Advanced Angiosarcoma and Other Soft Tissue Sarcomas
Brief Title: A Study of Axitinib in Patients With Advanced Angiosarcoma and Other Soft Tissue Sarcomas
Acronym: Axi-STS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other); Cancer Research UK (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH15195; 2008-006007-23 (EudraCT Number)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2019-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: advanced soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental): Patients will take axitinib tablets 5 mg by mouth twice daily continuously. There may be one dose reduction to 3mg twice daily.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Patients will take axitinib tablets 5 mg by mouth twice daily continuously. There may be one dose reduction to 3mg twice daily. A four week dosing period will be considered as 1 cycle of treatment. Axitinib treatment will be continued until disease progression, or the development of limiting toxicity.
  Other Names: AG-013736

SUMMARY:
The study objective is to evaluate the therapeutic activity, safety and tolerability of axitinib in patients with advanced/metastatic soft tissue sarcoma who are unsuitable for or have relapsed after standard chemotherapy. The therapeutic activity will be separately assessed in angiosarcoma, synovial sarcoma, leiomyosarcomas and other sarcomas.

DETAILED DESCRIPTION:
Soft tissue sarcomas are a heterogeneous group of rare malignancies that account for 0.72% of new malignancies and 0.65% of malignant deaths. Advanced sarcomas carry a poor prognosis. Angiogenesis is a hallmark of tumour growth, and there is increasing evidence that antiangiogenic drugs, including axitinib, can lead to tumour regression and improve patient survival in a variety of tumours.

Patients with angiosarcoma, synovial sarcoma, leiomyosarcoma and other sarcomas will be separately evaluated.

Patients will take axitinib 5mg tablets by mouth twice daily. This will be continued for 2 years or until disease progression, or development of limiting toxicity. In the event of severe toxicity, axitinib will be stopped until the toxicity has improved. Treatment may be interrupted for a maximum of 2 weeks. Following this, axitinib can be restarted at a lower dose of 3 mg twice daily. If the toxicity has not improved sufficiently, axitinib will be permanently stopped.

Patients will be monitored once weekly for the first month, then at 4 week intervals. Toxicity will be closely monitored. At each clinic visit, patients will have a physical examination and a routine blood test. A Chest x-ray, CT and/or MRI scans will be done before study entry, then every 12 weeks and at the end of treatment. Disease evaluation will be carried out 12 weeks after study entry, then every 12 weeks until disease progression. After disease progression, patients will be followed up every 3 months for survival. Patients will be followed up until death or a minimum follow up period of 1 year.

Patients will be enrolled from hospitals all over the UK.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed soft tissue sarcoma, including:

  * Angiosarcoma, including intermediate and malignant vascular tumours (WHO classification, 2002) and Kaposi's sarcoma.
  * Leiomyosarcoma, including uterine, skin or non organ origin.
  * Synovial sarcoma.
  * Other eligible subtypes of soft tissue sarcoma of Trojani intermediate or high grade, including fibroblastic, fibrohistiocytic, adipocytic, rhabdomyosarcoma, malignant peripheral nerve sheath, and not otherwise specified. See exclusion criteria for ineligible subtypes.
* Locally advanced or metastatic disease incurable by surgery or radiotherapy.
* Measurable disease according to RECIST criteria.
* Evidence of objective disease progression in the past 6 months, without anticancer treatment since progression.
* Patients ineligible for chemotherapy (eg. through age, clinical condition or patient refusal) or who have received no more than two prior chemotherapy regimens.
* Age >or = 16.
* WHO performance status 0, 1 or 2.
* At least 4 weeks from prior anticancer treatment (surgery, radiotherapy and systemic therapies) and full recovery from all their adverse effects.
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be < or = 140 mm Hg, and the baseline diastolic blood pressure readings must be < or = 90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Adequate physiological function:

  * renal : calculated or measured creatinine clearance > or = 50 ml/min using the Cockcroft-Gault formula (see appendix 5).
  * haematological: Absolute Neutrophil Count (ANC) > or = 1.5 x 109/L, platelets > or = 100 x 109/L, International Normalized Ratio (INR) < or = 1.2.
  * hepatic: bilirubin within normal range, AST and ALT < or = 3 x upper limit of normal.
  * cardiac: Left Ventricular Ejection Fraction (LVEF) measured by Echocardiogram or Multi Gated Acquisition Scan (MUGA) within normal range.
  * Urinary protein <2+ by urine dipstick. If dipstick is >2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours.
* Negative pregnancy test and agrees to comply with contraceptive measures
* Able to swallow oral medication.

Exclusion Criteria:

* Ineligible pathological subtypes including:

  * Osteosarcoma
  * Ewings/Primitive Neuroectodermal Tumour (PNET sarcomas)
  * Chondrosarcoma
  * Gastrointestinal stromal tumours (GIST)
  * Dermatofibrosarcoma protuberans (DFSP)
  * Malignant mesothelioma
  * Mixed mesodermal tumours of uterus
  * Known central nervous system metastases.
  * Age < 16.
  * Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, primidone, rifabutin, rifampicin, and St. John"s Wort).
* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, voriconazole, erythromycin, clarithromycin, ergot derivatives, indinavir, saquinavir, ritonavir, nelfinavir and lopinavir).
* Previous malignancies (except curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix or breast) within the past 3 years.
* Heart failure > or = New York Heart Association (NYHA) class II.
* History within the previous 6 months of any blood clots in the sputum or streaky haemoptysis that was persistent (> 2 weeks) or recurrent (> 3 episodes).
* Patients with cavitating lung metastases or any metastasis abutting or invading a major pulmonary blood vessel on baseline CT or MRI scan.
* History of bleeding diathesis or coagulopathy within 12 months of study entry
* Any of the following within the 12 months prior to trial drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, deep vein thrombosis or pulmonary embolism.
* Therapeutic dose warfarin. Low molecular weight heparin is permitted.
* Regular treatment with antiplatelet medication, including aspirin >325 mg/day or NSAIDs
* History of malabsorption or major gastrointestinal tract resection likely to affect trial drug absorption.
* Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use two effective contraception measures during the period of therapy which should be continued for 4 weeks after the last dose of trial therapy. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy which should be continued for 4 weeks after the last dose of trial therapy . The definition of effective contraception will be based on the judgment of the Investigator or designee.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2016-06-11 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 12 weeks after starting treatment, defined according to the Response Evaluation Criteria In Solid Tumours(RECIST criteria) | 12 weeks after trial entry, the final analysis of the primary outcome measure will take place after all patients have been followed for a minimum of 12 weeks
  Disease will be assessed by CT or MRI scan 12 weeks after entry to trial and will be compared to disease measured by CT or MRI scan on entry to the trial or within 4 weeks prior to entry. Response at 12 weeks will be measured using RECIST criteria. Progression-free survival rate is measured as the number of patients who are alive and progression-free at 12 weeks divided by the total number of patients who received at least one cycle of treatment

SECONDARY OUTCOMES:
Tumour response rate (using RECIST criteria) | 12 weeks and final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Disease will be assessed at 12 weeks by CT or MRI scan and clinical photographs where indicated, and compared with disease measured at baseline. Response will be measured using RECIST criteria. Tumour response rate is defined as the number of patients who achieved a complete or partial response divided by the total number of patients who received at least one cycle of treatment.
Progression-free interval | final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Progression-free interval is defined as the time from trial entry to date when disease progression first observed where progression is defined in terms of RECIST criteria. Patients who die of disease without disease progression being recorded are defined as progression at date of death. Those that die of other causes are censored at date of death and those who are alive with no recorded progression at time of analysis are censored at date last seen alive and progression-free.
Progression-free survival time | final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Progression-free survival time is defined in the same way as progression-free interval except that all deaths, whatever the cause, are included as events in the analysis.
Overall survival time | final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Survival time is measured from trial entry to death from any cause or to date last seen alive for those patients who are still alive at the time of analysis.
Change in performance status | final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Changes in performance status from baseline according to the World Health Organisation (WHO) performance status scale.
Toxicity rate | final analysis of all outcome measures will take place after all patients have been followed up for a minimum of 1 year.
  Adverse events will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Toxicity rate is defined as the number of patients experiencing at least one grade 3, 4 or serious adverse reaction divided by the total number of patients who started treatment

CONTACTS AND LOCATIONS:
Overall Officials: Penella Woll, BMedSci, Principal Investigator — Weston Park Hospital, Sheffield, UK
Locations (13):
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Bristol Haematology & Oncology Centre, Bristol
  - St. James's Hospital, Leeds
  - Royal Marsden Hospital, London
  - Royal Marsden, London
  - University College London Hospitals, London
  - Christies, Manchester
  - Clatterbridge Centre for Oncology, Metropolitan Borough of Wirral
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Penella Woll, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No